CLINICAL TRIAL: NCT03692975
Title: Hippocampal Microstructure Assessed by a New MRI Sequence and Episodic Memory at the Early Stage of Multiple Sclerosis: Comparison Between Patients After a Clinically Isolated Syndrome (CIS) and Controls
Brief Title: MRI Hippocampal Microstructure and Episodic Memory in Early Multiple Sclerosis
Acronym: Micro-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2017/30
Record Dates: First submitted 2018-08-07; First posted 2018-10-02 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis
Keywords: Clinically Isolated Syndrome; NODDI; Hippocampus; episodic memory function; dentate gyrus; MRI
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIS patients (Experimental): Clinically isolated neurological syndrome (CIS) compatible with a demyelinating inflammatory episode within the central nervous system, potentially suggestive of multiple sclerosis (MS) whatever the mode of presentation
  Interventions: Other: Clinical assessment; Other: Neuropsychological evaluation; Other: Psychological evaluation; Device: MRI Evaluation
- Control (Active Comparator): 50 Healthy controls
  Interventions: Other: Neuropsychological evaluation; Other: Psychological evaluation; Device: MRI Evaluation

INTERVENTIONS:
Other: Clinical assessment — Expanded Disability Status Scale (EDSS), ambulation test and Multiple Sclerosis functional composite (MSFC). Medications will be recorded.
  Arms: CIS patients
Other: Neuropsychological evaluation — cognitive tests exploring episodic memories, information processing speed, attention/concentration and working memory.
Other: Psychological evaluation — included questionnaires for depression, anxiety, fatigue, cognitive complaint and reserve
Device: MRI Evaluation — Diffusion including NODDI, 3DT1 with and without gadolinium, 3D-FLAIR before and after gadolinium infusion, 3D White Matter nulled-MPRAGE, 3D Double-Inversion recovery sequences-weighted imaging and Resting state functional MRI

SUMMARY:
Clinically isolated syndrome (CIS) can evolve into multiple sclerosis. In CIS patients, episodic memory is frequently impaired. Memory disorders could be preceded by microstructural abnormalities without visible atrophy in hippocampus. A recent MRI imaging of diffusion called NODDI (Neurite Orientation Dispersion and Density Imaging) can measure specifically microstructural abnormalities and map the axons in the white matter (WM) and dendrites in the grey matter (GM). The aim of this study is to evaluate microstructural abnormalities in the dentate gyrus of the hippocampus in CIS patients compared to controls.

DETAILED DESCRIPTION:
Cognitive deficiencies could occur after a first clinical event of the central nervous system suggestive of MS called clinically isolated syndrome (CIS). Cognitive impairment concerned several cognitive domains including episodic memory, attention, working memory and executive functions. It is recognized the negative impact of cognitive impairment on quality of life and vocational status in patients living with MS. Slowness of information processing speed is the main cognitive dysfunction observed in MS seen at the earliest stage of the disease. Recently an international group of MS experts has explain IPS and episodic memory as the minimal cognitive assessment in patients with MS. Visuospatial and verbal episodic memory deficits have been observed in 18 to 28% of patients assessed after a CIS.

Memory disorders could be preceded by microstructural abnormalities without visible atrophy in hippocampus. A recent MRI imaging of diffusion called NODDI (Neurite Orientation Dispersion and Density Imaging) can measure specifically microstructural abnormalities and map the axons in white matter and dendrite in the gray matter. No study has used the NODDI in CIS patients and very few studies have been conducted in MS.

The hypothesis is that the dentate gyrus is the anatomical substrate of early episodic memory dysfunction in patients included after a CIS.

The identification of predictive MRI biomarker of memory impairment would be a useful and clinically relevant prognostic marker at the early stage of MS. This biomarker could contribute to determine the prognosis of the disease and could help for the monitoring of the patients in clinical practice and clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* - PATIENTS:

  * Men and Women,
  * Age 18-60 years,
  * Native French language,
  * Clinically isolated neurological syndrome (CIS) compatible with a demyelinating inflammatory episode within the central nervous system, potentially beginning multiple sclerosis (MS) whatever the mode of presentation,
  * Between 60 and 180 days from the onset,
  * At least two clinically silent lesions on their T2-weighted brain or spinal MRI scan with a size of least 3 mm, at least one of which being cerebral, ovoid, or periventricular,
  * Willing to participate and to sign informed consent.
* - HEALTHY CONTROLS

  * Men and Women,
  * Age 18-60years,
  * Native French language,
  * Willing to participate and to sign informed consent.

Exclusion Criteria:

* - PATIENTS:

  * Prior documented neurological episode suggestive of MS,
  * History of neurological disease and/or other neurological diseases,
  * Psychiatric diseases,
  * Known chronic systemic diseases as judged by the investigator,
  * Alcohol or other addiction to toxic,
  * Disabling visual or motor problems preventing participation to neuropsychological assessments,
  * Acquisition disorders : Dyslexia, Dysphasia, Dyscalculia and dyspraxia,
  * Dosage change, stop or start of hypnotic or anxiolytic or antidepressive treatment less than 30 days,
  * Contra-indication to MRI (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body, claustrophobia),
  * Steroid treatment less than one month (be taken orally or by infusion) at the dosage of 500mg daily,
  * Illiteracy, is unable to count or to read,
  * Pregnant or breastfeeding women,
  * Patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent).
* - HEALTHY CONTROLS

  * History of neurological disease and/or neurological diseases,
  * Psychiatric diseases,
  * Known chronic systemic diseases as judged by the investigator,
  * Alcohol or other addiction to toxic,
  * Acquisition disorders: Dyslexia, Dysphasia, Dyscalculia and dyspraxia,
  * Known cognitive impairment or Prior neuropsychological testing with the same tests less than one year,
  * Hypnotic or anxiolytic or antidepressive treatment,
  * Steroid treatment less than one month (be taken orally or by infusion) at the dosage of 500mg daily,
  * Contra-indication to MRI (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body, claustrophobia) or refusing MRI,
  * Illiteracy, unable to count or to read,
  * Pregnant or breastfeeding women,
  * Patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Index of orientation-dispersion (IOD) | At baseline (day 0)
  This parameter is measured in the dentate gyrus of hippocampus from NODDI imaging blind to the nature of the patient's group (CIS patients and controls).
Index of Neurite density (ND) | At baseline (day 0)
  This parameter is measured in the dentate gyrus of hippocampus from NODDI imaging blind to the nature of the patient's group (CIS patients and controls).

SECONDARY OUTCOMES:
Diffusion parameters : Index of orientation-dispersion | At baseline (day 0)
  This parameter is measured in thalamus and cerebellum from NODDI imaging blind to the nature of the patient's group (CIS patients and controls).
Diffusion parameters : Neurite density | At baseline (day 0)
  This parameter is measured in thalamus and cerebellum from NODDI imaging blind to the nature of the patient's group (CIS patients and controls).
Diffusion parameters : Fractional Anisotropy | At baseline (day 0)
  This parameter is measured in dentate gyrus of hippocampus, thalamus and cerebellum from diffusion imaging blind to the nature of the patient's group (CIS patients and controls).
Diffusion parameters : Mean diffusivity | At baseline (day 0)
  This parameter is measured in dentate gyrus of hippocampus, thalamus and cerebellum from diffusion imaging blind to the nature of the patient's group (CIS patients and controls).
Atrophy parameters | At baseline (day 0)
  Normalized total brain volume and normalized total WM and total GM volumes and in hippocampus, thalamus and cerebellum from 3D-T1, 3D-DIR, 3D-WMn-MPRAGE in CIS patients and controls in double-blind.
Lesion volume | At baseline (day 0)
  Normalized volume of lesions double-blind measured by a semi-automatic method based on 3 D Fast Fluid-attenuated inversion-recuperation (3D-FLAIR) and 3 D Double Inversion Recovery (3D-DIR) in whole brain and in the hippocampus, thalamus and cerebellum.
Inflammatory activity | At baseline (day 0)
  The inflammatory activity will be the number of T1-gadolinium enhancing lesions in whole brain and in the hippocampus, thalamus and cerebellum.
Connectivity | At baseline (day 0)
  The seed-based connectivity is measured between hippocampus and others cerebral regions (Thalamus, cerebellum…) from Diffusion Tensor Imaging (DTI) and resting state functional imaging.
Verbal episodic memory test | At baseline (day 0)
  California Verbal Learning Test-Second version (CVLT-II)
Visual episodic memory score | At baseline (day 0)
  Brief Visual Memory Test-Revised (BVMT-R) and Memonic Similarity Task (MST) : visuospatial memory tests (2 scores pour BVMT-R, 3 scores pour MST)
Information processing speed and attention score | At baseline (day 0)
  Computerized Speed Cognitive Test (CSCT) and TAP
Working memory score | At baseline (day 0)
  Paced-Auditory-Serial-Addition-Test (PASAT) and span

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie RUET, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Eric FRISON, MD, PhD, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de neurologie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No